CLINICAL TRIAL: NCT02628249
Title: Application of Indicator Amino Acid Oxidation Method to Investigate the Rate-limiting Amino Acids in Endurance Trained Athlete
Brief Title: Rate-limiting Amino Acids in Endurance-trained Athlete
Acronym: EA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Moore, Assistant professaor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IAAO-EA
Record Dates: First submitted 2015-12-07; First posted 2015-12-11 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Increased Metabolic Requirement; Healthy
MeSH Terms: interventions — Amino Acids; Amino Acids, Essential

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Base protein (Experimental): 0.8 g/kg/d of protein provided as crystalline amino acid made after egg protein.
  Interventions: Dietary Supplement: Base protein
- Sufficient protein (Experimental): 1.75 g/kg/d protein provided as crystalline amino acid made after egg protein.
  Interventions: Dietary Supplement: Sufficient protein
- Base + BCAA (Experimental): Base protein intake + Branched chain amino acids
  Interventions: Dietary Supplement: Base protein; Dietary Supplement: Branched chain amino acids
- Base + EAA (Experimental): Base protein intake + essential amino acids.
  Interventions: Dietary Supplement: Base protein; Dietary Supplement: Essential amino acids
- Base + NEAA (Experimental): Base protein intake + non essential amino acids
  Interventions: Dietary Supplement: Base protein; Dietary Supplement: Non essential amino acids

INTERVENTIONS:
Dietary Supplement: Base protein — 0.8 g/kg/d of protein provided as crystalline amino acid modeled after egg protein
  Arms: Base + BCAA; Base + EAA; Base + NEAA; Base protein
Dietary Supplement: Sufficient protein — 1.75 g/kg/d protein provided as crystalline amino acid modeled after egg protein.
  Arms: Sufficient protein
Dietary Supplement: Branched chain amino acids — Branched chain amino acids modeled after egg protein.
  Arms: Base + BCAA
Dietary Supplement: Essential amino acids — Essential amino acids modeled after egg protein.
  Arms: Base + EAA
Dietary Supplement: Non essential amino acids — Non essential amino acids modeled after egg protein.
  Arms: Base + NEAA

SUMMARY:
Protein requirements in individuals who participate in endurance-based exercise training have been suggested to be greater than the current recommended dietary allowance (RDA).

The biological value of protein depends on the amino acid composition. As liebig's law of the minimum, the protein synthesis is limited due to the lack of single rate limiting amino acid. In this case, the first rate limiting amino acid determines protein intakes to maximize the protein synthesis. Adding a small amount of rate-limiting amino acid to the diet improves the biological value of its protein diet.

The indicator amino acid oxidation (IAAO) method has clarified the individual amino acid requirement in children, normal healthy adult and clinical populations. however, the IAAO method has never been utilized for determining the first rate limiting amino acid.

Therefore, the purpose of this study is to address of IAAO method to be applied for determining the rate-limiting amino acid in endurance athlete.

ELIGIBILITY:
Gender: Male

Age limit: Minimum age 18 years - Maximum age 35 years

Accepts Healthy Volunteers : yes

Inclusion Criteria:

* Endurance-trained participants who regularly more than 40 km/week
* Ability to perform the exercise stimulus (20 km run) on metabolic trial.

Exclusion Criteria:

* Inability to meet health and physical activity guidelines according to the physical activity readiness questionnaire (PAR-Q+)
* Inability to adhere to any of the protocol guidelines (i.e. alcohol, caffeine consumption)
* Regular tobacco use
* Illicit drug use

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
13CO2 (carbon dioxide) excretion rate (μmol/kg/h) | At 8 hours after the end of exercise
  8 hours after exercise followed by ingesting 13C-labelled phenylalanine and one of 5 different amount of amino acids intake, 13CO2 excretion rate is determined by multiplying the enrichment of 13CO2 in breath measured by Mass spectrometry and CO2 production rate measured by metabolic cart.

SECONDARY OUTCOMES:
[13C]phenylalanine oxidation rate (μmol/kg/h) | at 8 hours after the end of exercise
  8 hours after exercise followed by ingesting 13C-labelled phenylalanine and one of 5 different amount of amino acids intake, 13CO2 excretion rate is determined dividing 13CO2 excretion rate by urinary enrichment of 13C-phenylalanine in breath measured by Mass spectrometry, and CO2 production rate measured by metabolic cart.

REFERENCES:
- [Derived] Kato H, Suzuki K, Bannai M, Moore DR. Branched-Chain Amino Acids Are the Primary Limiting Amino Acids in the Diets of Endurance-Trained Men after a Bout of Prolonged Exercise. J Nutr. 2018 Jun 1;148(6):925-931. doi: 10.1093/jn/nxy048. PMID 29746639